CLINICAL TRIAL: NCT02690038
Title: Feasibility and Safety of Immunoglobulin (Ig) Prophylactic Treatment in COPD Patients With Frequent Exacerbations: A Pilot Study
Brief Title: Ig PRx in AECOPD: Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: CSL Behring (Industry); Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20150925 / 20160077-01H
Record Dates: First submitted 2016-02-10; First posted 2016-02-24 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: AECOPD; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Immunoglobulins, Intravenous; Octagam; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Arm 1: Treatment (Experimental): Baseline Ig < 7g/L group - Intravenous immunoglobulin (IVIG) 0.8 g/kg will be given within 12 hours after randomization during hospital admission and then every 4 weeks for 44 weeks (total 48 weeks).
  Baseline Ig > or = 7 g/L group - Intravenous immunoglobulin (IVIG) 0.5 g/kg will be given within 12 hours after randomization during hospital admission and then every 4 weeks for 44 weeks (total 48 weeks).
  Interventions: Drug: Intravenous immunoglobulin (IVIG)
- Intervention Arm 2: Control (Active Comparator): Baseline Ig < 7g/L group - Normal Saline (0.9% NaCl) 8 mL/kg will be given within 12 hours after randomization during hospital admission and then every 4 weeks for 44 weeks (total 48 weeks).
  Baseline Ig > or = 7 g/L group - Normal Saline (0.9% NaCl) 5 mL/kg will be given within 12 hours after randomization during hospital admission and then every 4 weeks for 44 weeks (total 48 weeks).
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Intravenous immunoglobulin (IVIG) — Baseline Ig < 7g/L group - Intravenous immunoglobulin (IVIG) 0.8 g/kg will be given within 12 hours after randomization.
  Baseline Ig > or = 7 g/L group - Intravenous immunoglobulin (IVIG) 0.5 g/kg will be given within 12 hours after randomization
  Other Names: Gamunex; CBS IGIV-nex; Privigen; Octagam
  Arms: Intervention Arm 1: Treatment
Drug: Normal Saline — Baseline Ig < 7g/L group - Normal Saline (0.9% NaCl) 8 mL/kg will be given within 12 hours after randomization.
  Baseline Ig > or = 7 g/L group - Normal Saline (0.9% NaCl) 5 mL/kg will be given within 12 hours after randomization
  Other Names: Saline; Sodium Chloride
  Arms: Intervention Arm 2: Control

SUMMARY:
This study will look at immunoglobulin (Ig) treatment in hospitalized chronic obstructive lung disease (COPD) patients with frequent exacerbations.

This is a Phase II, pilot randomized double blind control study, meaning this study will help assess if this research can be expanded to evaluate Ig treatment in patients with COPD. Ig treatment is a sterile solution of human immunoglobulin proteins given intravenously (in the vein). Immunoglobulins are part of the immune system and help the body fight infections. Participants will be assigned to either receiving the Ig treatment or normal saline as a control product every 4 weeks for 12 months.

Participants will continue on current standard therapy as determined by their treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult patient with AECOPD (clinically dominant AECOPD in the case of multiple co-morbidities eg. absence of overt lobar pneumonia or acute congestive heart failure or alternate diagnosis such as acute coronary syndrome or pulmonary embolism)
* Diagnosis of severe COPD (post bronchodilator FEV1 <50%, FEV1/FVC ratio <0.7) made by standard spirometry within previous 12 months or within three days of admission if previous PFT data is not available
* Age >40 years
* >10 pack year smoking history
* At least one COPD exacerbation in the previous 12 months before enrollment, defined by having had documented inpatient or outpatient treatment by physician with antibiotics and/or prednisone for physician diagnosed COPD exacerbation
* Expected to live > 12 months

Exclusion Criteria:

* Known severe hypersensitivity to immunoglobulin or its components (anaphylaxis)
* Underlying malignancy (including chronic lymphocytic leukemia)
* History of hematopoietic stem cell transplant or solid organ transplant
* Current treatment with a biological therapy for other conditions
* Concomitant significant immunodeficiency or on immunosuppressive treatment other than for COPD
* Alpha-1 antitrypsin deficiency
* Significant proteinuria (dipstick proteinuria ≥ 3+ or known urinary protein loss ≥ 2 g/day or nephrotic syndrome) and/or has acute renal failure and/or severe renal impairment (creatinine more than 2.5 times the upper limit of normal and/or on dialysis)
* IgA deficiency (IgA <0.1 g/L)
* Immunoglobulin therapy in the last 12 months or on current Ig therapy or have a clinical indication for Ig replacement therapy (www.nacblood.ca/resources/guidelines/IVIG.html)
* Obesity (BMI ≥35 kg/m²)
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09; Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Recruitment | 52 weeks
  Average number of patients being recruited per month. The study meets primary outcome if at least 4 patients can be recruited per month on average.
Adherence and protocol compliance | 104 weeks
  Number and percentage of recruited patients adhere to the allocated treatment and protocol. We aim to achieve 80% adherence rate which is defined as at least 80% of patients adhere to 80% of allocated treatment and protocol

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE | 104 weeks
  This will be assessed by documentation of adverse events in patients treated with Ig treatment versus control
Tolerability of treatment | 104 weeks
  The proportion of patients able to complete the treatment in the experimental arm during the study period versus in the control arm
Efficacy trend: Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) rates | 104 weeks
  AECOPD will be ascertained by monthly follow-up phone calls as well as questionnaires during study visits to detect inpatient/outpatient treatment for exacerbations.
Efficacy trend: Health status | 104 weeks
  measured by the validated St. George Respiratory Questionnaire
Efficacy trend: Quality of life | 104 weeks
  validated quality of life measurement tool - EuroWol EQ-5D-5L
Efficacy trend: % predicted FEV1 | 104 weeks
  FEV1 value will be measured using a hand held spirometer. FEV1 value will be recorded in Litres (L) and reported as a percent of their predicted value (using the NHANES III reference standards for predicted values
Efficacy trend: FEV1/FVC | 104 weeks
  FVC will be measured using a hand held spirometer, and will be recorded in Litres (L). Ratio of FEV1 and FVC will be reported.
Efficacy trend: Health services use | 104 weeks
  Number of non-study physician visits, emergency department (ED) and hospital admissions over the twelve-month study period.
Efficacy trend: Health care system cost | 104 weeks
  we will take the perspective of healthcare system and will measure the cost of health services use and an intervention. Intervention cost includes medication, staff, and equipment cost.

CONTACTS AND LOCATIONS:
Overall Officials: Juthaporn Cowan, MD, PhD, FRCPC, Principal Investigator — Associate Scientist
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cowan J, Gaudet L, Mulpuru S, Corrales-Medina V, Hawken S, Cameron C, Aaron SD, Cameron DW. A Retrospective Longitudinal Within-Subject Risk Interval Analysis of Immunoglobulin Treatment for Recurrent Acute Exacerbation of Chronic Obstructive Pulmonary Disease. PLoS One. 2015 Nov 11;10(11):e0142205. doi: 10.1371/journal.pone.0142205. eCollection 2015. PMID 26558756
- [Background] Niewoehner DE, Rice K, Cote C, Paulson D, Cooper JA Jr, Korducki L, Cassino C, Kesten S. Prevention of exacerbations of chronic obstructive pulmonary disease with tiotropium, a once-daily inhaled anticholinergic bronchodilator: a randomized trial. Ann Intern Med. 2005 Sep 6;143(5):317-26. doi: 10.7326/0003-4819-143-5-200509060-00007. PMID 16144890
- [Background] Hurst JR, Vestbo J, Anzueto A, Locantore N, Mullerova H, Tal-Singer R, Miller B, Lomas DA, Agusti A, Macnee W, Calverley P, Rennard S, Wouters EF, Wedzicha JA; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Susceptibility to exacerbation in chronic obstructive pulmonary disease. N Engl J Med. 2010 Sep 16;363(12):1128-38. doi: 10.1056/NEJMoa0909883. PMID 20843247
- [Background] Seemungal TA, Donaldson GC, Paul EA, Bestall JC, Jeffries DJ, Wedzicha JA. Effect of exacerbation on quality of life in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 May;157(5 Pt 1):1418-22. doi: 10.1164/ajrccm.157.5.9709032. PMID 9603117
- [Background] Toy EL, Gallagher KF, Stanley EL, Swensen AR, Duh MS. The economic impact of exacerbations of chronic obstructive pulmonary disease and exacerbation definition: a review. COPD. 2010 Jun;7(3):214-28. doi: 10.3109/15412555.2010.481697. PMID 20486821
- [Background] Mullerova H, Maselli DJ, Locantore N, Vestbo J, Hurst JR, Wedzicha JA, Bakke P, Agusti A, Anzueto A. Hospitalized exacerbations of COPD: risk factors and outcomes in the ECLIPSE cohort. Chest. 2015 Apr;147(4):999-1007. doi: 10.1378/chest.14-0655. PMID 25356881
- [Background] Baker CL, Zou KH, Su J. Risk assessment of readmissions following an initial COPD-related hospitalization. Int J Chron Obstruct Pulmon Dis. 2013;8:551-9. doi: 10.2147/COPD.S51507. Epub 2013 Nov 12. PMID 24348031
- [Background] Albert RK, Connett J, Bailey WC, Casaburi R, Cooper JA Jr, Criner GJ, Curtis JL, Dransfield MT, Han MK, Lazarus SC, Make B, Marchetti N, Martinez FJ, Madinger NE, McEvoy C, Niewoehner DE, Porsasz J, Price CS, Reilly J, Scanlon PD, Sciurba FC, Scharf SM, Washko GR, Woodruff PG, Anthonisen NR; COPD Clinical Research Network. Azithromycin for prevention of exacerbations of COPD. N Engl J Med. 2011 Aug 25;365(8):689-98. doi: 10.1056/NEJMoa1104623. PMID 21864166
- [Background] Zheng JP, Wen FQ, Bai CX, Wan HY, Kang J, Chen P, Yao WZ, Ma LJ, Li X, Raiteri L, Sardina M, Gao Y, Wang BS, Zhong NS; PANTHEON study group. Twice daily N-acetylcysteine 600 mg for exacerbations of chronic obstructive pulmonary disease (PANTHEON): a randomised, double-blind placebo-controlled trial. Lancet Respir Med. 2014 Mar;2(3):187-94. doi: 10.1016/S2213-2600(13)70286-8. Epub 2014 Jan 30. PMID 24621680
- [Background] Calverley PM, Rabe KF, Goehring UM, Kristiansen S, Fabbri LM, Martinez FJ; M2-124 and M2-125 study groups. Roflumilast in symptomatic chronic obstructive pulmonary disease: two randomised clinical trials. Lancet. 2009 Aug 29;374(9691):685-94. doi: 10.1016/S0140-6736(09)61255-1. PMID 19716960
- [Background] Han MK, Martinez FJ. Pharmacotherapeutic approaches to preventing acute exacerbations of chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2011 Aug;8(4):356-62. doi: 10.1513/pats.201102-016RM. PMID 21816992
- [Background] Brightling CE, Bleecker ER, Panettieri RA Jr, Bafadhel M, She D, Ward CK, Xu X, Birrell C, van der Merwe R. Benralizumab for chronic obstructive pulmonary disease and sputum eosinophilia: a randomised, double-blind, placebo-controlled, phase 2a study. Lancet Respir Med. 2014 Nov;2(11):891-901. doi: 10.1016/S2213-2600(14)70187-0. Epub 2014 Sep 7. PMID 25208464
- [Background] Kawano T, Matsuse H, Obase Y, Kondo Y, Machida I, Tomari S, Mitsuta K, Fukushima C, Shimoda T, Kohno S. Hypogammaglobulinemia in steroid-dependent asthmatics correlates with the daily dose of oral prednisolone. Int Arch Allergy Immunol. 2002 Jul;128(3):240-3. doi: 10.1159/000064258. PMID 12119507
- [Background] Yip NH, Lederer DJ, Kawut SM, Wilt JS, D'Ovidio F, Wang Y, Dwyer E, Sonett JR, Arcasoy SM. Immunoglobulin G levels before and after lung transplantation. Am J Respir Crit Care Med. 2006 Apr 15;173(8):917-21. doi: 10.1164/rccm.200510-1609OC. Epub 2006 Jan 6. PMID 16399990
- [Background] Kazatchkine MD, Kaveri SV. Immunomodulation of autoimmune and inflammatory diseases with intravenous immune globulin. N Engl J Med. 2001 Sep 6;345(10):747-55. doi: 10.1056/NEJMra993360. No abstract available. PMID 11547745
- [Background] Ochsenbein AF, Fehr T, Lutz C, Suter M, Brombacher F, Hengartner H, Zinkernagel RM. Control of early viral and bacterial distribution and disease by natural antibodies. Science. 1999 Dec 10;286(5447):2156-9. doi: 10.1126/science.286.5447.2156. PMID 10591647
- [Background] Gelfand EW. Intravenous immune globulin in autoimmune and inflammatory diseases. N Engl J Med. 2012 Nov 22;367(21):2015-25. doi: 10.1056/NEJMra1009433. No abstract available. PMID 23171098
- [Background] Gilardin L, Bayry J, Kaveri SV. Intravenous immunoglobulin as clinical immune-modulating therapy. CMAJ. 2015 Mar 3;187(4):257-264. doi: 10.1503/cmaj.130375. Epub 2015 Feb 9. No abstract available. PMID 25667260
- [Background] Sabroe I, Postma D, Heijink I, Dockrell DH. The yin and the yang of immunosuppression with inhaled corticosteroids. Thorax. 2013 Dec;68(12):1085-7. doi: 10.1136/thoraxjnl-2013-203773. Epub 2013 Aug 8. No abstract available. PMID 23929790
- [Background] Fedor ME, Rubinstein A. Effects of long-term low-dose corticosteroid therapy on humoral immunity. Ann Allergy Asthma Immunol. 2006 Jul;97(1):113-6. doi: 10.1016/S1081-1206(10)61380-4. PMID 16892792
- [Background] Kaveri SV, Maddur MS, Hegde P, Lacroix-Desmazes S, Bayry J. Intravenous immunoglobulins in immunodeficiencies: more than mere replacement therapy. Clin Exp Immunol. 2011 Jun;164 Suppl 2(Suppl 2):2-5. doi: 10.1111/j.1365-2249.2011.04387.x. PMID 21466545
- [Background] Orange JS, Grossman WJ, Navickis RJ, Wilkes MM. Impact of trough IgG on pneumonia incidence in primary immunodeficiency: A meta-analysis of clinical studies. Clin Immunol. 2010 Oct;137(1):21-30. doi: 10.1016/j.clim.2010.06.012. Epub 2010 Aug 1. PMID 20675197
- [Derived] Cowan J, Mulpuru S, Abdallah SJ, Chopra A, Purssell A, McGuinty M, Alvarez GG, Giulivi A, Corrales-Medina V, MacFadden D, Boyle L, Hasimja D, Thavorn K, Mallick R, Aaron SD, Cameron DW. A Randomized Double-Blind Placebo-Control Feasibility Trial of Immunoglobulin Treatment for Prevention of Recurrent Acute Exacerbations of COPD. Int J Chron Obstruct Pulmon Dis. 2021 Dec 3;16:3275-3284. doi: 10.2147/COPD.S338849. eCollection 2021. PMID 34887657
- [Derived] Cowan J, Mulpuru S, Aaron S, Alvarez G, Giulivi A, Corrales-Medina V, Thiruganasambandamoorthy V, Thavorn K, Mallick R, Cameron DW. Study protocol: a randomized, double-blind, parallel, two-arm, placebo control trial investigating the feasibility and safety of immunoglobulin treatment in COPD patients for prevention of frequent recurrent exacerbations. Pilot Feasibility Stud. 2018 Aug 11;4:135. doi: 10.1186/s40814-018-0327-z. eCollection 2018. PMID 30116551
- See also: Microsoft Word - OLA Final Report June 21 - document.doc. — https://lungontario.ca/
- See also: Chronic Obstructive Pulmonary Disease (COPD) Fact Sheet - American Lung Association. — http://www.lung.org/lung-disease/copd/resources/facts-figures/COPD-Fact-Sheet.html#Burden.
- See also: Chronic Obstructive Pulmonary Disease (COPD) Evidentiary Framework - Health Quality Ontario (HQO). — http://www.hqontario.ca/evidence/publications-and-ohtac-recommendations/ontario-health-technology-assessment-series/chronic-obstructive-pulmonary-disease-copd-evidentiary-framework
- See also: GOLD_Pocket_2017_Feb18.pdf — https://goldcopd.org/wp-content/uploads/2016/12/wms-GOLD-2017-Pocket-Guide.pdf
- See also: Intravenous immunoglobulin enhances the killing activity and autophagy of neutrophils isolated from immunocompromised patients against multidrug-re... — http://www.ncbi.nlm.nih.gov/pubmed/26119690.